CLINICAL TRIAL: NCT03204331
Title: SPIRIT 2: An International Phase 3 Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study to Evaluate Relugolix Administered With and Without Low-Dose Estradiol and Norethindrone Acetate in Women With Endometriosis-Associated Pain
Brief Title: SPIRIT 2: Efficacy and Safety Study of Relugolix in Women With Endometriosis-Associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MVT-601-3102; 2017-001632-19 (EudraCT Number)
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Endometriosis Related Pain
Keywords: Endometriosis; Pain; Dysmenorrhea
MeSH Terms: conditions — Endometriosis; Pain; Dysmenorrhea | interventions — relugolix; estradiol, norethindrone drug combination; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relugolix plus E2/NETA (Group A) (Experimental): Relugolix co-administered with E2/NETA for 24 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate
- Relugolix plus Delayed E2/NETA (Group B) (Experimental): Relugolix co-administered with E2/NETA placebo for 12 weeks, followed by relugolix co-administered with E2/NETA for 12 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate; Drug: Estradiol/norethindrone acetate placebo
- Placebo (Group C) (Placebo Comparator): Relugolix placebo co-administered with E2/NETA placebo for 24 weeks.
  Interventions: Drug: Estradiol/norethindrone acetate placebo; Drug: Relugolix placebo

INTERVENTIONS:
Drug: Relugolix — Relugolix 40-mg tablet administered orally once daily.
  Other Names: TAK-385; MVT-601
  Arms: Relugolix plus Delayed E2/NETA (Group B); Relugolix plus E2/NETA (Group A)
Drug: Estradiol/norethindrone acetate — Capsule containing co-formulated tablet of E2 (1.0 mg)/NETA (0.5 mg) administered orally once daily.
  Other Names: E2/NETA
  Arms: Relugolix plus Delayed E2/NETA (Group B); Relugolix plus E2/NETA (Group A)
Drug: Estradiol/norethindrone acetate placebo — E2 (0 mg)/NETA (0 mg) placebo capsule administered orally once daily and designed to match the E2/NETA capsule in size, shape, color, and odor.
  Arms: Placebo (Group C); Relugolix plus Delayed E2/NETA (Group B)
Drug: Relugolix placebo — Relugolix (0 mg) placebo tablet administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor.
  Arms: Placebo (Group C)

SUMMARY:
The purpose of this study is to determine the benefit and safety of relugolix 40 milligrams (mg) once daily, co-administered with low-dose estradiol (E2) and norethindrone acetate (NETA) compared with placebo for 24 weeks, on dysmenorrhea and on nonmenstrual pelvic pain.

DETAILED DESCRIPTION:
This study is an international phase 3 randomized, double-blind, placebo-controlled efficacy and safety study to evaluate 24 weeks of oral, once-daily relugolix (40 mg) co-administered with either 12 or 24 weeks of low-dose E2 (1.0 mg) and NETA (0.5 mg), compared with placebo.

Approximately 600 women with endometriosis-associated pain were enrolled and randomized 1:1:1 to Group A - relugolix plus low-dose hormonal add-back therapy, Group B - relugolix monotherapy for 12 weeks followed by co-administration with low-dose hormonal add-back therapy, or Group C - placebo (N = 200 per group).

Eligible participants were randomized on Baseline Day 1 to Treatment Group A, B, or C, in the double-blind period.

Eligible participants, including those randomized to placebo, were offered the opportunity to enroll in an 80-week open label extension study where participants received relugolix co-administered with low-dose E2 and NETA. Participants who did not enroll into the extension study had a Follow-Up visit approximately 30 days after the participant's last dose of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is a premenopausal female aged 18 to 50 years old (inclusive) on the day of signing of the informed consent form.
2. Has agreed to use only study-specified analgesic medications during the study and is not known to be intolerant to these.
3. Has a diagnosis of endometriosis and has had, within 10 years prior to signing the informed consent form, surgical or direct visualization and/or histopathologic confirmation of endometriosis, for example, during a laparoscopy or laparotomy.
4. During the Run-In Period (35 to 70 days prior to treatment period) has a dysmenorrhea NRS score ≥ 4.0 on at least 2 days and

   1. Mean NMPP NRS score ≥ 2.5, or
   2. Mean NMPP NRS score ≥ 1.25 and NMPP NRS score ≥ 5.0 on ≥ 4 days.

Key Exclusion Criteria:

1. Has a history of chronic pelvic pain that is not caused by endometriosis.
2. Has any chronic pain or frequently recurring pain condition, other than endometriosis that is treated with opioids or requires analgesics for ≥ 7 days per month.
3. Has had surgical procedures for treatment of endometriosis within the 3 months prior to the Screening visit.
4. Has a history of or currently has osteoporosis or other metabolic bone disease.
5. Has a clinically significant gynecologic condition, other than endometriosis, identified during Screening or Run-In period transvaginal ultrasound or endometrial biopsy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 623 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage Of Participants Who Meet The Dysmenorrhea Responder Criteria At Week 24 Or End Of Treatment (EOT) | Week 24 or EOT
  Assessed using a Numerical Rating Scale (NRS) score (11-point scale) for pain recorded daily in an electronic diary (e-Diary). The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Percentage Of Participants Who Meet The Non-Menstrual Pelvic Pain (NMPP) Responder Criteria At Week 24 Or EOT | Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary. The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.

SECONDARY OUTCOMES:
Change From Baseline In The Endometriosis Health Profile (EHP)-30 Pain Score At Week 24 | Baseline, Week 24
  Assessed using the Pain Domain of the EHP-30 questionnaire.
Change From Baseline In Dysmenorrhea NRS Score At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change From Baseline In NMPP NRS Score At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change From Baseline In Overall Pelvic Pain NRS Score At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change From Baseline In Dyspareunia NRS Scores At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using an NRS score (11-point scale) for dyspareunia recorded daily in an e-Diary.
Percentage Of Participants Who Are Not Using Opioids For Endometriosis-associated Pain At Week 24 Or EOT | Week 24 or EOT
  Assessed based on usage of protocol-specified opioids for endometriosis-associated pain recorded daily in an e-Diary.
Change From Baseline In Analgesic Use For Endometriosis-associated Pain Based On Mean Pill Count At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed based on usage of protocol-specified analgesic for endometriosis-associated pain recorded daily in an e-Diary.
Percentage Of Participants Who Have A Reduction Of At Least 20 Points In The EHP-30 Pain Domain From Baseline To Week 24 | Baseline to Week 24
  Assessed using the pain domain of the EHP-30 questionnaire.
Dysmenorrhea Responder Rate By Month | Baseline to Week 24
  The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
NMPP Responder Rate By Month | Baseline to Week 24
  The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Change In Dysmenorrhea NRS Score By Month | Baseline to Week 24
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change In NMPP NRS Score By Month | Baseline to Week 24
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change In Overall Pelvic Pain NRS Score By Month | Baseline to Week 24
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change In Dyspareunia NRS Score By Month | Baseline to Week 24
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary.
Change From Baseline In Ibuprofen Use At Week 24 Or EOT | Baseline, Week 24
  Assessed using ibuprofen pill counts for endometriosis-associated pain recorded daily in an e-Diary.
Change From Baseline In Opioid Use At Week 24 Or EOT | Baseline, Week 24
  Assessed using opioid pill counts for endometriosis-associated pain recorded daily in an e-Diary.
Change From Baseline In The Mean Dysmenorrhea Functional Impairment At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using the subject modified Biberoglu and Behrman 5-point scale for dysmenorrhea recorded daily in an e-Diary.
Change From Baseline In The Mean NMPP Functional Impairment At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using the subject modified Biberoglu and Behrman 4-point scale for pelvic pain recorded daily in an e-Diary.
Change From Baseline In The Mean Dyspareunia Functional Impairment At Week 24 Or EOT | Baseline, Week 24 or EOT
  Assessed using the subject modified Biberoglu and Behrman 5-point scale for dyspareunia recorded daily in an e-Diary.
Change From Baseline In Patient Global Assessment (PGA) For Dysmenorrhea Symptom Severity At Week 24 | Baseline, Week 24
  The PGA for dysmenorrhea is a 1-item questionnaire designed to assess participants' impression of the severity of pain during their menstrual cycle.
Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA For Dysmenorrhea At Week 24 | Week 24
  The PGA for dysmenorrhea is a 1-item questionnaire designed to assess participants' impression of the severity of pain during their menstrual cycle.
Change From Baseline In PGA For NMPP Symptom Severity At Week 24 | Baseline, Week 24
  The PGA for NMPP is a 1-item questionnaire designed to assess participants' impression of the severity of pain when they are not menstruating.
Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA For NMPP At Week 24 | Week 24
  The PGA for NMPP is a 1-item questionnaire designed to assess participants' impression of the severity of pain when they are not menstruating.
Change From Baseline In PGA For Pain Severity At Week 24 | Baseline, Week 24
  The PGA for pain severity is a 1-item questionnaire designed to assess participants' impression of how their pain affected their usual activities.
Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA For Pain Severity At Week 24 | Week 24
  The PGA for pain severity is a 1-item questionnaire designed to assess participants' impression of how their pain affected their usual activities.
Change From Baseline In PGA For Function At Week 24 | Baseline, Week 24
  The PGA for function is a 1-item questionnaire designed to assess participants' impression of how their pain affected their usual activities.
Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA For Function At Week 24 | Week 24
  The PGA for function is a 1-item questionnaire designed to assess participants' impression of how their pain affected their usual activities.
Percentage Of Participants Who Are "Better" Or "Much Better" On The Patient Global Impression Of Change (PGIC) For Dysmenorrhea At Week 24 | Week 24
  The PGIC for dysmenorrhea is a 1-item questionnaire designed to assess participants' impression of change in the severity of pain during their menstrual cycle.
Percentage Of Participants Who Are "Better" Or "Much Better" On The PGIC For NMPP At Week 24 | Week 24
  The PGIC for NMPP is a 1-item questionnaire designed to assess participants' impression of change in the severity of pain during their menstrual cycle.
Percentage Of Participants Who Are "Better" Or "Much Better" On The PGIC For Dyspareunia At Week 24 | Week 24
  The PGIC for dyspareunia is a 1-item questionnaire designed to assess participants' impression of change in the severity of pain during sexual intercourse.
Change From Baseline In The Non-Pain Of The EHP-30 Domains At Week 24 | Baseline, Week 24
  Assessed using the non-pain domains (Control and Powerlessness, Social Support, Emotional Well-Being, and Self-Image) of the EHP-30 questionnaire.
Change From Baseline In The EHP-30 Scale Total Score At Week 24 | Baseline, Week 24
  Assessed using the total score of the EHP-30 questionnaire.
Change From Baseline In The EHP Work Domain Score At Week 24 | Baseline, Week 24
  The EHP Work domain is a 5-item questionnaire that assesses impact of pain on ability to work.
Categorical Change From Baseline In Quality Of Life Assessed By European Quality Of Life Five Dimension Five Level (EQ-5D-5L) Questionnaire At Week 24 | Baseline, Week 24
  The EQ-5D-5L is a 5-item questionnaire designed to assess quality of life.
Change From Baseline To Week 24 In EQ-5D-5L Visual Analogue Scale Score At Week 24 | Baseline, Week 24
  The EQ-5D-5L is a 5-item questionnaire designed to assess quality of life.
Percentage Of Participants Who Meet The Dysmenorrhea Responder Criteria At Week 24 Or EOT For Relugolix Plus Delayed E2/NETA | Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary. The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Percentage Of Participants Who Meet The NMPP Responder Criteria At Week 24 Or EOT For Relugolix Plus Delayed E2/NETA | Week 24 or EOT
  Assessed using an NRS score (11-point scale) for pain recorded daily in an e-Diary. The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Change From Baseline In The EHP-30 Pain Score At Week 24 For Relugolix Plus Delayed E2/NETA | Baseline, Week 24
  Assessed using the Pain Domain of the EHP-30 questionnaire.
Percentage Of Participants Who Have A Reduction Of At Least 20 Points In The EHP-30 Pain Domain From Baseline To Week 24 For Relugolix Plus Delayed E2/NETA | Baseline to Week 24
  Assessed using the pain domain of the EHP-30 questionnaire.
Percentage Change From Baseline In Bone Mineral Density At The Lumbar Spine (L1-L4) At Week 12 | Baseline, Week 12
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Percentage Change From Baseline In Bone Mineral Density At Lumbar Spine (L1-L4), Femoral Neck, And Total Hip At Week 24 | Baseline, Week 24
  Assessed by DXA scan.
Percentage Of Participants Experiencing Vasomotor Symptoms At Week 12 Between Group A And B | Week 12
Change From Baseline In Serum Concentrations Of Luteinizing Hormone, Follicle Stimulating Hormone, Estradiol, And Progesterone | Baseline, Week 24
  Blood samples will be collected from participants for hormonal measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (76):
- United States (39):
  - Andalusia, Andalusia, Alabama
  - Washington DC, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - Deland, DeLand, Florida
  - Hialeah, Hialeah, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - Port St. Lucie, Port Saint Lucie, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Park Ridge, Park Ridge, Illinois
  - Lafayette, Lafayette, Indiana
  - Covington, Covington, Louisiana
  - Marrero, Marrero, Louisiana
  - Towson, Towson, Maryland
  - Saginaw, Saginaw, Michigan
  - St. Louis, St Louis, Missouri
  - Omaha, Omaha, Nebraska
  - Albuquerque, Albuquerque, New Mexico
  - New York, New York, New York
  - New Bern, New Bern, North Carolina
  - Akron, Akron, Ohio
  - Columbus, Columbus, Ohio
  - Franklin, Franklin, Ohio
  - Columbia, Columbia, South Carolina
  - Spartanburg, Spartanburg, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Beaumont, Beaumont, Texas
  - Corpus Christi, Corpus Christi, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Houston, Houston, Texas
  - Irving, Irving, Texas
  - San Antonio, San Antonio, Texas
  - Sugar Land, Sugar Land, Texas
  - Pleasant Grove, Pleasant Grove, Utah
  - Salt Lake City, Salt Lake City, Utah
  - Virginia Beach, Virginia Beach, Virginia
- Australia (5):
  - Sydney, Sydney, New South Wales
  - Wollongong, Wollongong, New South Wales
  - Sherwood, Sherwood, Queensland
  - Adelaide, Adelaide, South Australia
  - Nedlands, Nedlands, Western Australia
- Brazil (5):
  - Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Porto Alegre, Porto Alegre, São Paulo
  - São Bernardo do Campo, São Bernardo do Campo, São Paulo
  - São Paulo, São Paulo, São Paulo
- Santiago, Santiago, Chile
- Czechia (4):
  - Tábor, Tábor, Jihormoravsky KRAJ
  - Písek, Písek, Jihočeský kraj
  - Praha 2, Prague, Prague
  - Ceské Budejovice, České Budějovice
- Tbilisi, Tbilisi, Borjomi, Georgia
- Italy (5):
  - Monserrato, Monserrato, Cagliari
  - Catanzaro, Catanzaro
  - Napoli, Napoli
  - Pavia, Pavia
  - Roma, Roma
- New Zealand (5):
  - Birkenhead, Birkenhead, Auckland
  - Remuera, Remuera, Auckland
  - Tauranga, Tauranga, Bay of Plenty
  - Palmerston North, Palmerston North, Manawatu-Wanganui
  - Christchurch, Christchurch
- Poland (7):
  - Poznan, Poznan, Greater Poland Voivodeship
  - Lublin, Lublin, Lublin Voivodeship
  - Warszawa, Warsaw, Masovian Voivodeship
  - Bialystok, Bialystok, Podlaskie Voivodeship
  - Białystok, Bialystok, Podlaskie Voivodeship
  - Katowice, Katowice, Silesian Voivodeship
  - Lodz, Lodz, Łódź Voivodeship
- Romania (3):
  - București, Bucharest, București
  - Brasov, Brasov
  - Bucuresti, Bucharest
- Malmö, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giudice LC, As-Sanie S, Arjona Ferreira JC, Becker CM, Abrao MS, Lessey BA, Dynowski K, Wilk K, Li Y, Mathur V, Wagman RB, Johnson NP. A Plain Language Summary to learn about relugolix combination therapy for the treatment of pain associated with endometriosis. Pain Manag. 2023 Nov;13(11):631-640. doi: 10.2217/pmt-2023-0052. Epub 2023 Nov 20. PMID 37982388
- [Derived] Hunsche E, Gauthier M, Witherspoon B, Rakov V, Agarwal SK. Endometriosis Symptoms and Their Impacts on the Daily Lives of US Women: Results from an Interview Study. Int J Womens Health. 2023 Jun 1;15:893-904. doi: 10.2147/IJWH.S409733. eCollection 2023. PMID 37283994
- [Derived] Giudice LC, As-Sanie S, Arjona Ferreira JC, Becker CM, Abrao MS, Lessey BA, Brown E, Dynowski K, Wilk K, Li Y, Mathur V, Warsi QA, Wagman RB, Johnson NP. Once daily oral relugolix combination therapy versus placebo in patients with endometriosis-associated pain: two replicate phase 3, randomised, double-blind, studies (SPIRIT 1 and 2). Lancet. 2022 Jun 18;399(10343):2267-2279. doi: 10.1016/S0140-6736(22)00622-5. PMID 35717987